CLINICAL TRIAL: NCT06102317
Title: The Effects of Smartphone-assisted Nursing Care Used for Mothers of Children With Cerebral Palsy Who Receive Home Healthcare Services on the Care Burden, Coping With Stress, and Quality of Life of Mothers
Brief Title: the Use of Smart Mobile Application in Mothers With Cerebral Palsy Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr. Behcet Uz Children's Hospital (Other)
Responsible Party: Principal Investigator, ÖKKEŞ KISA, The Effects of Smartphone-assisted Nursing Care Used for Mothers of Children With Cerebral Palsy Who Receive Home Healthcare Services on the Care Burden, Coping With Stress, and Quality of Life of Mothers, Dr. Behcet Uz Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Behcet-OKISA-001
Record Dates: First submitted 2023-10-08; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Cerebral Palsy
Keywords: "Cerebral Palsy"; "Quality of Life"; "Caregiver Burden"; "Smartphone"
MeSH Terms: conditions — Cerebral Palsy; Caregiver Burden

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): In the study, mobile application will be installed on the phones of the mothers in the initiative group and individual information will be provided about how the patients will use the smartphone application. . Information will be provided to patients for subsequent follow-ups. After the application is started to be used, notifications of the applications developed in Smart Mobile for the disease management process will be made to the mothers of the Initiative Group every two weeks for six months. In addition, the Initiative Group will continue to receive standard care practices such as examinations, examinations, tests, treatment, medical care and rehabilitation offered by the Home Health Services unit.
  Interventions: Other: nursing consultancy with smartphone support
- control group (No Intervention): No attempts will be made to the control group. The control group will continue to receive the standard care practices offered by the Home Health Services unit.

INTERVENTIONS:
Other: nursing consultancy with smartphone support — In the study, mobile application will be installed on the phones of the mothers in the initiative group and individual information will be provided about how the patients will use the smartphone application. . Information will be provided to patients for subsequent follow-ups. After the application is started to be used, notifications of the applications developed in Smart Mobile for the disease management process will be made to the mothers of the Initiative Group every two weeks for six months. In addition, the Initiative Group will continue to receive standard care practices such as examinations, examinations, tests, treatment, medical care and rehabilitation offered by the Home Health Services unit.
  Arms: Intervention group

SUMMARY:
There are studies in the literature aimed at supporting parents who care for children who have Cerebral Palsy. Among these, the study conducted on the use of mobile applications in supporting parents has attracted attention in recent years. When the studies on supporting parents were examined, it was found in one study that a mobile application designed for caregivers enabled parents to support their children's nutrition, bathing, toileting, playing, carrying, and movement training. As a result of this study, it was reported that the knowledge and skills of caregivers regarding the care of their children increased. It was emphasized in another study that mobile medicine applications that are developed for children who have disabilities such as Cerebral Palsy must have a drug list, drug name, drug reminder module, drug registration section, and additional characteristics. In a randomized controlled study, it was reported that a web-based daycare program designed for the children of mothers who had children with CP increased the quality of life of the mothers. In another study, it was explained to caregivers of children who had Cerebral Palsy that the application facilitated the daily care of children anytime and anywhere in a training module consisting of a mobile application with information about CP, nutrition, toilet, bath, transportation, games, and medication reminder modules. Studies conducted on the use of technology-based (telehealth, mobile applications, web-based education) healthcare service delivery, education, and consultancy services in supporting families in Turkey are limited. The present study aimed to reduce the care burden and stress of parents of children who had Cerebral Palsy and improve their quality of life with the mobile application developed with the support of nurses.

The purpose of the present study is to examine the effects of smartphone-supported nursing consultancy applied to mothers of children who have Cerebral Palsy receiving home healthcare services on their care burden, coping with stress, and quality of life

DETAILED DESCRIPTION:
Study Question In the present study, an answer will be sought to the question "Does the smartphone-supported nursing consultancy used by the mothers of children with Cerebral Palsy who receive home healthcare and are registered at S.B.U. Dr. Behçet Uz Pediatric Diseases and Surgery Training and Research Hospital Home Healthcare Services Unit located in Konak district of Izmir affect the mothers' care burden, coping with stress and quality of life?"

Hypotheses Hypothesis 1 (H1): There is a difference between the care burden scale scores of the Intervention and Control Group according to time (pre-test, 1st month after the intervention, 3rd month, 6th month).

Hypothesis 2 (H1): There is a difference between the quality of life scale scores of the Intervention and Control Group according to time (pre-test, 1st month after the intervention, 3rd month, 6th month).

Hypothesis 3 (H1): There is a difference between the stress scale scores of the Intervention and Control Group according to time (pre-test, 1st month after the intervention, 3rd month, 6th month).

Original value of the study Coordination between parents and healthcare professionals in pediatric home health services will be improved with the mobile application that will be developed as a result of the study and effective use of healthcare services will be ensured, contributing to the protection, development, and maintenance of healthcare.

There are many studies in the literature on the caregivers of children with Cerebral Palsy. However, no randomized controlled study was detected on the effects of mobile applications on care burden, stress, and quality of life. For this reason, it is expected to be an original study in this field and to contribute to the literature in planning future studies.

It is envisaged that nurses will reflect innovative and easy-to-access technological developments in nursing care, and the mobile application will form the basis for supportive studies based on mobile applications in the nursing care of parents.

Studies in the literature report that the quality of life of parents who had children with Cerebral Palsy decreased during the COVID-19 pandemic because of social distance and curfews, stress, their care burden increased, and they could not benefit from qualified healthcare services. For this reason, it is recommended to use telehealth services effectively during Covid-19 and in future epidemics/pandemics. For this reason, it is expected that parents' active participation and compliance with the treatment process will be easier because a smartphone-supported program will be used in the study and time will be saved in transportation to healthcare professionals.

It is expected that rapid insight into the existing evidence base will be provided at the intersection between policymakers, public healthcare staff, and other professionals who work in this field.

Study Design: The study will have a randomized controlled follow-up design with a pretest-posttest control group. The population of the study will consist of the mothers of 58 children diagnosed primarily with Cerebral Palsy among the 170 patients who receive home healthcare and are registered at S.B.U. Dr. Behçet Uz Pediatric Diseases and Surgery Training and Research Hospital Home Healthcare Services Unit located in the Konak district of Izmir. The study will be conducted in the home healthcare services of the hospital. The size of the study population was determined by the researcher from the results of the study titled "Retrospective evaluation of applications made to the home care services unit of a public hospital" with the decision of protocol 591 and 2021/12_09 to S.B.U. Dr. Behçet Uz Pediatric Diseases and Surgery Training and Research Hospital on 08.07.21.

A power analysis was performed to determine the sample size in the study by using the G*Power 3.1.9.7 program. The final tests of the total scores on the quality of life scale of study, which was previously conducted on a similar subject, were taken as a reference in determining the sample size of the study.

In the present study, it was envisaged to conduct a "t-test" (Experiment-Control) to determine whether the smartphone-supported nursing consultancy applied to mothers of children with Cerebral Palsy receiving home healthcare had an effect on the mothers' care burden, coping with stress, and quality of life. As a result of the analysis, the standardized effect size was found to be 0.93 at α=0.05 level (based on previous studies), and the minimum number of samples was determined to be 40 (20 in the first group and 20 in the second group) with a theoretical power of 0.95. It was emphasized in the literature that it must be taken into consideration that there will be a 20% case loss in randomized controlled studies; for this reason, the number of samples was determined as 48 (24 experimental; 24 control).

The Stratified Randomization Method will be used according to the gender and age of the children diagnosed with CP whom the mothers care for. The way randomization will be implemented based on the literature data, with the simple random sampling method because there of the lists of parents in the study previously conducted by the researcher to determine the population, the population was less than 1000 (N<1000) registered in the same unit, to ensure the homogeneity of the sample in the study. in this study, it was decided to use the Program "R 4.2.1" to strongly randomize and evenly distribute it to the intervention-control group at once.

Inclusion Criteria

1. Having a child with CP registered in the Home Healthcare Services Unit at S.B.U Dr. Behçet Uz Pediatric Diseases and Surgery Training and Research Hospital
2. Residing in the province of Izmir and at home
3. Having a primary diagnosis of Cerebral Palsy in the home health care file
4. The primary caregiver of the child is the mother
5. The mother does not have any communication or mental problems
6. The mother's ability to read and write in Turkish
7. Having an Android or IOS-based smartphone
8. Voluntary participation in the study

Exclusion Criteria

1. Children who were residing in the Ministry of Family and Social Policies Services.

Study Variables

The independent variable of the study: Status of receiving smartphone-supported nursing consultancy.

The dependent variable of the study: Zarit Care Burden Scale score, Parental Stress Index score, and Quality of Life Scale score.

Place and Time of Study The study will be conducted at S.B.U. Dr. Behçet Uz Pediatric Diseases and Surgery Training and Research Hospital Home Healthcare Services Unit located in the Konak district of Izmir. The study is planned to be conducted between 01 February 2024 and 31 July 2024. The pilot application of the smartphone application is planned between 01 february 2024 and 31 January 2024.

Data Collection A telephone conversation will be made with the mothers registered to the Home Healthcare Services Unit and meet the inclusion criteria and the necessary information will be given about the study during the data collection. The forms to be used in the pre-test will be collected from the mothers in the intervention and control groups with the face-to-face interview method by going to the homes of the mothers who agree to participate in the study, taking into account the necessary COVID-19 pandemic measures. A mobile application will be installed on the phones of the mothers in the intervention group and individual information will be given to the patients about how to use the smartphone application during these meetings and participants will be informed about follow-ups. After the application is started to be used, Intervention Group mothers will be notified of the applications developed for smart mobiles for the disease management process every two weeks for six months. Also, the Intervention Group will continue to receive standard care practices such as examination, analysis, treatment, medical care, and rehabilitation offered by the Home Health Services Unit.

No intervention will be made to the Control Group, which will continue to receive standard care practices provided by the Home Healthcare Services Unit.

The Smartphone Application for Parents of Children who have Primary Cerebral Palsy For the Intervention Group, the healthcare service needs of families who have children with Cerebral Palsy will be determined by examining them in line with the literature data. These nursing needs will be designed by a consulting company that specializes in the application. The content evaluation of the designed smartphone application will be made with the DISCERN Measurement Tool. Specialists in the field will be asked to fill out the DISCERN Measurement Tool and their opinions will be evaluated with the Kendall Coefficient of Concordance, which is an analysis method used to evaluate inter-rater concordance. Kendall is shown with "W". Kendall W can range from "0" (no concordance) to "1" (full concordance). As this value approaches "1", it indicates a good level of concordance among specialists. Then, a pilot study will be conducted to evaluate the effectiveness of the smartphone application and to identify the deficiencies, by taking institutional permission from 10% of the sample and testing it on mothers of children who are diagnosed with Cerebral Palsy in one of the private rehabilitation centers. The smartphone application will be finalized in line with the feedback that will be obtained from the pilot application. The content of the smartphone application will be created according to the literature data under the following headings.

1. Information on Cerebral Palsy
2. Medication reminder
3. Parental self-care plan
4. Exercise module
5. Fever management
6. Communication panel to ask questions to the specialist
7. Parent-Peer interaction

Data analysis The SPSS 22.0 Package program will be used to analyze the study data. The data will be evaluated statistically at a 95% Confidence Interval and a significance level of p<0.05. Numbers and percentage distributions will be used in the analysis of the data for sociodemographic characteristics. Parametric and nonparametric tests will be used after analyzing the suitability of the quantitative data for normal distribution.

ELIGIBILITY:
Inclusion Criteria:

1. Having a child with CP registered in the Home Healthcare Services Unit at S.B.U Dr. Behçet Uz Pediatric Diseases and Surgery Training and Research Hospital
2. Residing in the province of Izmir and at home
3. Having a primary diagnosis of Cerebral Palsy in the home health care file
4. The primary caregiver of the child is the mother
5. The mother does not have any communication or mental problems
6. The mother's ability to read and write in Turkish
7. Having an Android or IOS-based smartphone
8. Voluntary participation in the study

Exclusion Criteria:

* 1. Children who were residing in the Ministry of Family and Social Policies Services.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
the effect of nurse-assisted telephone application on quality of life, stress and care burden in mothers with cerebral palsy children | 1 month
  the change in the total scores of the smartphone mobile application applied nurse-assisted to the mothers in the intervention group on the stress, care burden and quality of life scale in the mothers in the intervention group in the study conducted at the end of 4 weeks

SECONDARY OUTCOMES:
the effect of nurse-assisted telephone application on quality of life, stress and care burden in mothers with cerebral palsy children | 3 month
  the change in the total scores of the smartphone mobile application applied nurse-assisted to the mothers in the intervention group on the stress, care burden and quality of life scale in the mothers in the intervention group in the study conducted at the end of 12 weeks

OTHER OUTCOMES:
the effect of nurse-assisted telephone application on quality of life, stress and care burden in mothers with cerebral palsy children | 6 month
  the change in the total scores of the smartphone mobile application applied nurse-assisted to the mothers in the intervention group on the stress, care burden and quality of life scale in the mothers in the intervention group in the study conducted at the end of 24 weeks

IPD SHARING:
Plan to Share IPD: No